CLINICAL TRIAL: NCT00022516
Title: Low-dose Cytotoxics as "Anti-angiogenesis Treatment" Following Adjuvant Induction Chemotherapy for Patients With ER-negative and PgR-negative Breast Cancer
Brief Title: Low-dose Oral Cyclophosphamide and Methotrexate Maintenance for Hormone Receptor-negative Early Breast Cancer
Acronym: 22-00
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068827; IBCSG-22-00 (Other: IBCSG); 2005-005666-36 (EudraCT Number); EU-20119 (Registry Identifier: NCI Liaison Office, Brussels)
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IB breast cancer; estrogen receptor-negative breast cancer; progesterone receptor-negative breast cancer; triple-negative breast cancer; low-dose maintenance chemotherapy; stroma; angiogenesis
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Cyclophosphamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No-CM (No Intervention): No further chemotherapy following standard adjuvant chemotherapy.
- CM-Maintenance (Experimental): 12-month CM-maintenance regimen (C, cyclophosphamide 50 mg/day orally continuously and M, methotrexate 2.5 mg twice/day orally days 1 and 2 of every week for 1 year)
  Interventions: Drug: Cyclophosphamide; Drug: Methotrexate

INTERVENTIONS:
Drug: Cyclophosphamide — 50 mg/day orally continuously for 1 year
  Other Names: Endoxan; Cytoxan
  Arms: CM-Maintenance
Drug: Methotrexate — 2.5 mg twice/day orally days 1 and 2 of every week for 1 year
  Other Names: Trexall
  Arms: CM-Maintenance

SUMMARY:
This randomized, phase III trial was designed to test the efficacy of a low-dose chemotherapy-maintenance regimen, hypothesized to have anti-angiogenic activity, administered following standard chemotherapy in patients with early breast cancer whose tumors are hormone receptor negative.

DETAILED DESCRIPTION:
PURPOSE:

* Evaluate a low-dose cyclophosphamide and methotrexate chemotherapy-maintenance regimen in early breast cancer.
* Compare the disease-free survival, overall survival, and systemic disease-free survival of patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.

OUTLINE:

This is a randomized, open-label, multicenter study. Patients are stratified according to participating center, menopausal status (pre vs post), and approved induction chemotherapy (anthracycline and cyclophosphamide vs other agents). Treatment duration is 12 months of low-dose chemotherapy-maintenance regimen (CM-maintenance) vs no chemotherapy-maintenance regimen (no-CM) following standard adjuvant chemotherapy. Patients are randomized to one of two treatment arms. Patients are followed every 6 months for 5 years, and yearly follow-up thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I, II, or III breast cancer

  * T1-3, N0-2, M0

    * Patients with sentinel node biopsy positive disease must have undergone axillary dissection
    * Tumor must be confined to the breast without detected metastases elsewhere
  * T4 disease with minimal dermal invasion allowed
  * No T4 disease with ulceration of skin, infiltration of skin (except pathologically minimal dermal involvement), peau d'orange, or inflammatory breast cancer
* No bilateral breast cancer (except in situ carcinoma) or suspicious mass in opposite breast that has not been proven benign
* No distant metastases

  * No skeletal pain of unknown cause, elevated alkaline phosphatase, or bone scan showing hot spots that cannot be ruled out as metastases by x-ray, MRI, and/or CT
* Must have undergone prior total mastectomy OR breast-conserving procedure (e.g., lumpectomy, quadrantectomy, or partial mastectomy with negative margins) with radiotherapy planned

  * Patients must begin or have begun an approved induction chemotherapy regimen within 8 weeks after definitive surgery
* Negative surgical margins
* Axillary clearance with at least 6 lymph nodes examined OR negative sentinel node biopsy
* Known HER2 status by immunohistochemistry or fluorescence in situ hybridization
* Hormone receptor status:

  * Estrogen and progesterone receptor negative

    * Less than 10% positive tumor cells by immunohistochemistry

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Not specified

Menopausal status:

* Premenopausal, defined as less than 6 months since last menstrual period (LMP) AND no prior bilateral ovariectomy AND not on estrogen replacement (OR under age 50) OR
* Postmenopausal, defined as prior bilateral ovariectomy OR more than 12 months since LMP without prior hysterectomy (OR age 50 and over)

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 3,000/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* See Disease Characteristics
* Bilirubin less than 2.0 mg/dL
* ALT less than 1.5 times upper limit of normal OR AST less than 60 IU/L

Renal:

* Creatinine less than 1.2 mg/dL

Other:

* Not pregnant or lactating within the past 6 months
* Fertile patients must use effective barrier contraception
* No other prior or concurrent malignancy except adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or contralateral or ipsilateral in situ breast carcinoma
* No psychiatric or addictive disorders that would preclude study
* No non-malignant systemic disease that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior trastuzumab (Herceptin) allowed

Chemotherapy:

* See Disease Characteristics
* No prior adjuvant or neoadjuvant chemotherapy for breast cancer

Endocrine therapy:

* No prior endocrine therapy for breast cancer or prevention
* No prior tamoxifen or raloxifene for breast cancer

Radiotherapy:

* No prior radiotherapy for breast cancer except primary irradiation

Surgery:

* See Disease Characteristics

Other:

* No prior preventative therapy for breast cancer

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1086 (Actual)
Dates: Start 2000-11; Primary Completion 2015-01 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Colleoni, MD, Study Chair — European Institute of Oncology
Locations (36):
- Australia (6):
  - Tweed Heads Hospital, Tweed Heads, New South Wales
  - Queen Elizabeth Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Maroondah Hospital, East Ringwood, Victoria
  - Murray Valley Private Hospital and Cancer Treatment Centre, Wodonga, Victoria
  - Christchurch Hospital, Christchurch
- CHU Liege - Domaine Universitaire du Sart Tilman, Liège, Belgium
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Chile (5):
  - Fundacion Arturo Lopez Perez, Santiago
  - Centro de Estudios Oncologicos Santiago, Santiago
  - Hospital Clinico San Borja Arriaran, Santiago
  - Hospital Clinico Universidad de Chile, Santiago
  - Hospital Carlos Van Buren, Valparaíso
- National Institute of Oncology - Budapest, Budapest, Hungary
- Italy (10):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale degli Infermi - ASL 12, Biella
  - Ospedale Civile Ramazzini, Carpi
  - Ospedale Alessandro Manzoni, Lecco
  - Ospedale San Paolo, Milan
  - European Institute of Oncology, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Civile Rimini, Rimini
  - Ospedale Sant' Eugenio, Rome
  - Policlinico Universitario Udine, Udine
- University of Ibadan Health Center, Ibadan, Nigeria
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Institutul Oncologic - Universitatea de Medicina, Cluj-Napoca, Romania
- Sandton Oncology Centre, Johannesburg, South Africa
- Switzerland (8):
  - Kantonsspital Aarau, Aarau
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - FMH Onkologie/Haematologie, Rheinfelden
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Colleoni M, Gray KP, Gelber S, Lang I, Thurlimann B, Gianni L, Abdi EA, Gomez HL, Linderholm BK, Puglisi F, Tondini C, Kralidis E, Eniu A, Cagossi K, Rauch D, Chirgwin J, Gelber RD, Regan MM, Coates AS, Price KN, Viale G, Goldhirsch A. Low-Dose Oral Cyclophosphamide and Methotrexate Maintenance for Hormone Receptor-Negative Early Breast Cancer: International Breast Cancer Study Group Trial 22-00. J Clin Oncol. 2016 Oct 1;34(28):3400-8. doi: 10.1200/JCO.2015.65.6595. Epub 2016 Jun 20. PMID 27325862
- [Result] Pruneri G, Gray KP, Vingiani A, Viale G, Curigliano G, Criscitiello C, Lang I, Ruhstaller T, Gianni L, Goldhirsch A, Kammler R, Price KN, Cancello G, Munzone E, Gelber RD, Regan MM, Colleoni M. Tumor-infiltrating lymphocytes (TILs) are a powerful prognostic marker in patients with triple-negative breast cancer enrolled in the IBCSG phase III randomized clinical trial 22-00. Breast Cancer Res Treat. 2016 Jul;158(2):323-31. doi: 10.1007/s10549-016-3863-3. Epub 2016 Jul 2. PMID 27372069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1086 patients were randomized between November 2000 and December 2012.
Period: Overall Study
Arm/Group | No-CM | CM-Maintenance
Started | 542 | 544
Completed | 539 | 314
Not Completed | 3 | 230
Not completed — Adverse Event | 0 | 59
Not completed — Lack of Efficacy | 0 | 27
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 2 | 113
Not completed — Incomplete documentation | 0 | 27

BASELINE CHARACTERISTICS:
Population: Patients who started overall study
Groups:
- Total: Total of all reporting groups
Arm/Group | No-CM | CM-Maintenance | Total
Number analyzed (Participants) | 542 | 544 | 1086
Age, Continuous [Median (Full Range); unit: years] | 52 [28 to 80] | 52 [28 to 79] | 52 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 542 | 544 | 1086
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where disease-free survival is defined as the time from randomization to the first appearance of one of the following: invasive breast cancer recurrence at local, regional, or distant site, invasive contralateral breast cancer, second (non-breast) invasive cancer, or death without cancer event; or censored at date of last follow-up.
Time Frame: 5-year estimates, reported at a median follow-up of 6.9 years
Population: Intention to treat (N=1081 patients)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No-CM | CM-Maintenance
Number analyzed (Participants) | 539 | 542
percentage of participants | 74.7 [70.6 to 78.3] | 78.1 [74.2 to 81.6]
Statistical Analysis 1: Comparison: No-CM vs CM-Maintenance; Test type: Superiority or Other; p = 0.14, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.6 to 1.06]

2. Secondary Outcome: Overall Survival
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where overall survival is defined as the time from randomization to death from any cause; or censored at date last known alive.
Time Frame: 5-year estimates, reported at a median follow-up of 6.9 years
Population: Intention to treat (N=1081 patients)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No-CM | CM-Maintenance
Number analyzed (Participants) | 539 | 542
percentage of participants | 85.0 [81.5 to 87.9] | 85 [81.5 to 88.0]
Statistical Analysis 1: Comparison: No-CM vs CM-Maintenance; Test type: Superiority or Other; p = 0.3570, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.65 to 1.17]

3. Secondary Outcome: Distant Recurrence-free Interval
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where distant recurrence-free Interval is defined as the time from randomization to invasive breast cancer recurrence at distant site, or invasive contralateral breast cancer; or censored at date of last follow up.
Time Frame: 5-year estimates, reported at a median follow-up of 6.9 years
Population: Intention-to-treat (N=1081 patients)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No-CM | CM-Maintenance
Number analyzed (Participants) | 539 | 542
percentage of participants | 83.5 [79.9 to 86.5] | 85.5 [79.9 to 86.5]
Statistical Analysis 1: Comparison: No-CM vs CM-Maintenance; Test type: Superiority or Other; p = 0.3178, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.62 to 1.17]

4. Secondary Outcome: Breast Cancer-free Interval
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where breast cancer-free interval is defined as the time from randomization to invasive breast cancer recurrence at local, regional, or distant site, or invasive contralateral breast cancer; or censored at date of last follow up.
Time Frame: 5-year estimates, reported at a median follow-up of 6.9 years
Population: Intention-to-treat (N=1081 patients)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No-CM | CM-Maintenance
Number analyzed (Participants) | 539 | 542
percentage of participants | 77.3 [73.3 to 80.7] | 81.0 [77.2 to 84.2]
Statistical Analysis 1: Comparison: No-CM vs CM-Maintenance; Test type: Superiority or Other; p = 0.06, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.6 to 1.01]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected every 3 months during the 12-month CM-maintenance chemotherapy treatment period.
Description: Only Grade 3 and higher AEs were collected among patients who initiated the experimental (CM-Maintenance) therapy (N=473) . AE data were NOT collected for patients who did not receive CM-maintenance therapy (No-CM)
Arm/Group | No-CM | CM-Maintenance
Serious Adverse Events (participants affected / at risk) | 0/0 | 11/473
Other Adverse Events (participants affected / at risk) | 0/0 | 58/473
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No-CM (N=0) | CM-Maintenance (N=473)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1
CNS hemorrhage (Nervous system disorders) | 0 (0) | 1
Elevated SGPT (Hepatobiliary disorders) | 0 (0) | 1
Neurologic-other (Nervous system disorders) | 0 (0) | 1
Ocular-other (Eye disorders) | 0 (0) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No-CM (N=0) | CM-Maintenance (N=473)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 8
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Arrhythmia-other (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1
Peripheral arterial ischemia (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Elevated GGT (Hepatobiliary disorders) | 0 | 1
Elevated SGOT (Hepatobiliary disorders) | 0 | 9
Elevated SGPT (Hepatobiliary disorders) | 0 | 32
Infection w/ unknown ANC (Infections and infestations) | 0 | 1
Infection w/o neutropenia (Infections and infestations) | 0 | 2
Infection w/ grade 3 or 4 neutropenia (Infections and infestations) | 0 | 1
Joint, muscle, bone-other (Musculoskeletal and connective tissue disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Neuropathy-sensory (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Abdominal pain (General disorders) | 0 | 1
Headache (General disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
This trial collected only Grade 3 or higher Adverse Events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No